CLINICAL TRIAL: NCT03053895
Title: Bedside Versus Operating Room Burr-Hole Drainage of Chronic Subdural Hematoma (DECIDE)
Acronym: DECIDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Saleh Almenawer, Neurosurgeon, Division of Neurosurgery, Principal Investigator, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19122016
Record Dates: First submitted 2016-12-26; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSDH Bedside twist drill technique (Experimental): For patients randomized to bedside drainage of Chronic Subdural Hematoma, the twist-drill procedure will be conducted at the patient's bedside using local anesthetic.
  Interventions: Procedure: CSDH - Bedside twist drill technique
- CSDH Operating Room Burr-hole technique (Active Comparator): For patients randomized to burr-hole drainage, the procedure will be performed in the operating room under local or general anesthesia based on the surgeon's and anesthesiologist's judgement of the clinical stability of the patient.
  Interventions: Procedure: CSDH - Operating Room Burr-hole technique

INTERVENTIONS:
Procedure: CSDH - Bedside twist drill technique — For patients randomized to bedside drainage of CSDH, the twist-drill procedure will be conducted at the patient's bedside using local anesthetic
  Arms: CSDH Bedside twist drill technique
Procedure: CSDH - Operating Room Burr-hole technique — For patients randomized to burr-hole drainage, the procedure will be performed in the operating room under local or general anesthesia based on the surgeon's and anesthesiologist's judgement of the clinical stability of the patient.
  Arms: CSDH Operating Room Burr-hole technique

SUMMARY:
DECIDE (Bedside versus Operating Room Burr-Hole DrainagE of ChronIc SubDural HEmatoma)

CSDH is an abnormal collection of blood between the layers of the brain causing brain tissue compression leading to neurological complications. One of the most common risk factors contributing to CSDH is head trauma, which is usually in the form of a minor head injury. Older individuals are at increased risk of CSDH due to brain atrophy that occurs with advancing age as well as their tendency to fall and sustain minor head traumas. Chronic alcoholics are also at increased risk as alcoholism also leads to brain atrophy, increased risk of falls, and liver failure which results in increased bleeding risk. Also many drugs used today like anticoagulants, antithrombotics, and antiplatelets for certain health conditions are other common risk factors for CSDH.

The overall goal of this multi-centered trial in the USA and Canada is to assess the surgical management of chronic subdural hematoma (CSDH) and to demonstrate the effectiveness of bedside drainage and its safety as it bypasses the perioperative risk associated with anesthetic especially among the elderly.

Adult patients with a clear indication for CSDH drainage will be randomly assigned to one of two procedures. One group will receive the twist drill procedure which can be performed at the bedside. The second group will undergo the burr-hole drainage procedure in the operating room usually under general anesthetic. Typically, the twist drill procedure can occur sooner as the operating room and Anesthetist are not required. Reoccurrence of the CSDH will be assessed over a period of 6 months following drainage. Timing of procedure, risk of infection, adverse side effects and neurological functioning will also be measured.

Over a 3 year study period, 486 eligible patients (243 patients per arm) will be enrolled. Patients > 18 years with confirmed diagnosis of symptomatic CSDH will be provided one of the two procedures and will be followed for study outcomes at 1, 3 and 6 months following the procedure.

Primary analysis will be to compare the surgical procedures, assessing the recurrence rate of CSDH within 6 months of initial CSDH drainage.

The ultimate goal of this study is to standardize bedside drainage as the treatment of choice for CSDH management.

This trial is important in the ongoing search for more efficient and safe intervention strategies.

DETAILED DESCRIPTION:
DECIDE (Bedside versus Operating Room Burr-Hole DrainagE of ChronIc SubDural HEmatoma)

Background and Significance: Chronic subdural hematoma (CSDH) is an abnormal collection of liquefied blood products between the dura and arachnoid membranes of the brain that may cause brain tissue compression and subsequent neurological sequelae. One of the most common risk factors contributing to CSDH is head trauma, which is usually in the form of a minor head injury. Older individuals are at increased risk of CSDH due to brain atrophy that occurs with advancing age as well as their tendency to fall and sustain minor head traumas. Chronic alcoholics are also at increased risk as alcoholism leads to globalized brain atrophy, increased risk of falls, and hepatogenic coagulopathy. Coagulopathies including the use of anticoagulants, antithrombotics, and antiplatelets for certain health conditions are other common risk factors for CSDH.

Study Aims: The primary aim of our study is to conduct a high-quality randomized trial to compare the safety and effectiveness of the bedside and operating room burr-hole drainage of CSDH. The main objective of this study is to demonstrate the effectiveness of bedside drainage and its safety as it bypasses the perioperative risk associated with anesthetic especially among the elderly.

The ultimate goal of this study is to standardize bedside drainage as the treatment of choice for CSDH management.

Primary Objective: To assess the efficacy of bedside drainage compared to operating room burr-hole evacuation for CSDH management by examining the hypothesis that bedside is associated with lower recurrence rate.

Secondary Objectives: To examine if the bedside drainage and the operating room burr-hole drainage are efficacious in terms of functional outcomes. To evaluate the hypothesis that bedside drainage is safer compared to the operating room burr-hole drainage by measuring mortality and morbidity.

Overall study design: Multi-centered pragmatic randomized controlled trial across North America (USA and Canada) comparing bedside drainage with operating room burr-hole drainage of CSDH.

Duration: Over a 3 year study period, each patient will be followed for 6 months to measure the study outcomes.

Study population: The study population will include 486 eligible patients >18 years of age with confirmed diagnosis of symptomatic CSDH (243 patients per arm).

Inclusion Criteria: Patients aged > 18 years presenting with symptomatic CSDH confirmed on diagnostic imaging, who are able to provide informed consent or have a legal representatives available if unable to do so.

Main intervention and comparator(s): Patients will be randomly assigned between the two arms of the study, bedside and operating room burr-hole drainage. For patients randomized to bedside drainage of CSDH, the twist-drill procedure will be conducted at the patient's bedside using local anesthetic. For patients randomized to burr-hole drainage, the procedure will be performed in the operating room under local or general anesthesia based on the surgeon's and anesthesiologist's judgement of the clinical stability of the patient. Randomization via www.randomize.net website will be stratified by center and by patient age in variable unspecified block sizes.

Follow-Up Post-Randomization: Patients randomized will be followed for study outcomes on days 1, 2, discharge, and months 1, 3 and 6.

Primary Outcome: The efficacy of comparative surgical procedures will be measured by the recurrence rate of CSDH within 6 months of initial CSDH drainage.

Secondary Functional Outcomes: Postoperative neurological and functional status of the patients will be measured using the Markwalder Grading System (MGS), Glasgow Outcome Score (GOS), and modified Rankin Scale (MRS).

Secondary Safety Outcomes: The safety of both procedures will be measured in terms of mortality and morbidity including surgical site infections, misplacement of postoperative subdural drain, tension pneumocephalus, new intracranial hemorrhage, and other medical complications.

Sample Size: Sample size estimation is based on a Chi-squared two-sided test of the null hypothesis that bedside drainage is not different from burr-hole drainage in reducing the proportion of patients who experience a hematoma recurrence within 6 months of the drainage procedure. Including for possible attrition rate of 10% a total of 486 patients (243 per arm) will be required to detect a difference in recurrence rates of 7% or a risk ratio of 0.36 (11% in the burr-hole group and 4% in the bedside drainage group), with a power of 80% and a level of significance set at alpha=0.05.

Primary Analysis: Primary analysis will be by intention-to-treat and data analyst will be blinded to participant allocation.

Interim Analyses: Interim analyses will be conducted upon recruitment of 25% of the expected sample size (122 patients) to assess recruitment rates, recurrence rates and safety outcomes.

This trial is important in the ongoing search for more efficient and safe intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >/= 18 years
* Presenting with symptomatic Chronic Subdural Hematoma confirmed on diagnostic imaging
* Able to provide informed consent or have a legal representatives available if unable to do so

Exclusion Criteria:

* Patients with acute or subacute subdural hematoma
* Patients with incidental or asymptomatic findings on CT; skull base, posterior fossa, or in the inter-hemispheric fissure Chronic Subdural Hematoma
* Patients with recurrent hematoma within 6 months of initial drainage
* Patients with Chronic Subdural Hematoma from previous intracranial surgery for different pathology Patients with subdural hygroma and non-hairline skull fracture over the Chronic Subdural Hematoma
* Patients with significant cognitive impairment or severe co-morbidity preventing improvement or follow-up
* Patients with hemorrhagic tendency that cannot be normalized
* Patients on anticoagulants, antithrombotics, or antiplatelets unless reversed or cleared - Patients who are unlikely to be available for a 6-month follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of Chronic Subdural Hematoma | 6 months

SECONDARY OUTCOMES:
Postoperative neurological and functional status - MGS | 6 Months
  Postoperative neurological and functional status using Markwalder Grading System
Postoperative neurological and functional status - GOS | 6 Months
  Postoperative neurological and functional status using Glasgow Outcome Score
Postoperative neurological and functional status - MRS | 6 Months
  Postoperative neurological and functional status using modified Rankin Scale
surgical site infection rate | 6 Months
  The safety of both procedures will be measured in terms of surgical site infections
safety - misplacement of postoperative subdural drain | 6 Months
  The safety of both procedures will be measured in terms of misplacement of postoperative subdural drain
new intracranial hemorrhage rate | 6 Months
  The safety of both procedures will be measured in terms of new intracranial hemorrhage
tension pneumocephalus | 6 Months
  The safety of both procedures will be measured in terms of tension pneumocephalus
mortality | 6 Months
  The safety of both procedures will be measured in terms of mortality
morbidity | 6 Months
  The safety of both procedures will be measured in terms of morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Almenawer, MD, Principal Investigator — Hamilton Health Sciences Corporation

IPD SHARING:
Plan to Share IPD: No